CLINICAL TRIAL: NCT03728712
Title: Quantitative Ventilation Lung Single-photon Emission Computed Tomography With CT Scan (Technegas SPECT/CT) to Assess Early Small Airway Disease in Smokers: a Pilot Study
Brief Title: Evaluation of Ventilation Homogeneity as a Marker of Small Airway Disease in Active Smokers
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Cyclomedica Australia PTY Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: 18.149
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Lung Function Testing; Cigarette Smoking; Single-photon Emission Computed Tomography (SPECT); Ventilation Homogeneity; Lung Disease Prevention
MeSH Terms: conditions — Cigarette Smoking | interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Never smokers: Participants with no history of cigarette smoking
  Interventions: Diagnostic Test: SPECT/CT
- Active smokers: Participants with an active history of cigarette smoking AND at least 10 pack-years total smoking history
  Interventions: Diagnostic Test: SPECT/CT

INTERVENTIONS:
Diagnostic Test: SPECT/CT — Technegas-Tc99m is approved by Health Canada for the evaluation of ventilation. Technegas will be prepared with a Technegas Generator (Cyclomedica) according to the manufacturer recommendations with a simmer phase and a burning phase. 95% ethanol will be used to wet the carbon crucible. The crucible will be loaded with 20-30 mCi of Tc99m. Tc99m has a physical half-life of 6 hours.
  Technegas will be administered to the patient within 10 minutes of its preparation, in a separate room than the scanning room. The inhalation technique will be rehearsed with the patient prior to the actual inhalation. The patient will be in supine position. A mouth piece and a nose clip will be used. The patient will be instructed to take 3 breaths of Technegas, starting after normal exhalation. A survey meter will be used to monitor the quality of the inhalation.

SUMMARY:
Ventilation heterogeneity is a hallmark feature of most obstructive pulmonary diseases. In particular, chronic obstructive pulmonary disease (COPD) is pathologically and physiologically characterized by small airway destruction and marked airway cellular inflammation, which result in prominent expiratory airflow limitation, air trapping, hyperinflation and abnormal gas exchange. COPD is strongly linked with the exposition to inhaled irritants, most notably tobacco smoke, and is as such a potentially preventable disease. COPD-related morbidity, mortality and social costs are high: in Canada, COPD is the main cause of hospital admission among all chronic diseases and is the fourth leading cause of death.

Diagnosis of COPD requires the objective demonstration of expiratory airflow limitation using spirometry. In the right clinical context, a post-bronchodilator forced vital capacity (FVC) / forced expiratory volume in 1 second (FEV1) ratio <0.70 is considered indicative of the presence of COPD, and therefore pulmonary function testing is required to make the diagnosis. However, the natural history of COPD represents a slowly-progressive continuum: active smokers that do not meet the criteria for COPD are still at risk of developing the disease. In fact, when compared to healthy non-smokers, active smokers without overt COPD can already show some pathological and clinical features of the disease. Notably, they report increased levels of resting dyspnea, chronic cough, lower exercise capacity, exercise-induced dynamic hyperinflation and marked airway inflammatory cellular infiltration, while conserving normal pulmonary function test values.

These findings highlight the negative, clinically-measurable effects of tobacco smoking on pulmonary function, but also the limitations of standard pulmonary function testing in identifying the presence of early, mild airway disease and quantifying physiological limitations in these subjects. As such, there is a need for a novel, simple and reliable method of quantifying airway disease in this population.

Quantitative lung ventilation single-photon emission computed tomography (SPECT) allows an objective quantification of the regional heterogeneity of ventilation in humans. The coefficient of variation (CV) of the distribution of a radioactive tracer, inhaled during the test, allows the generation of heterogeneity maps and density curves of small elements of the lung. These variables are sensitive to the presence of COPD, asthma, air trapping and are correlated to even slight anomalies in pulmonary function testing in otherwise healthy subjects. As such, SPECT could prove useful as an early marker of airway disease in active smokers at risk of developing COPD, but its use in this context has never been formally tested.

This pilot study addresses the question of whether lung SPECT could provide clinically relevant information on airway disease in active smokers without overt lung disease on pulmonary lung function testing.

ELIGIBILITY:
For Smokers group:

Inclusion Criteria:

* Active tobacco smoking of at least 10 cigarettes/day AND total smoking history of at least 15 pack-years.
* Normal lung function testing, defined as: FVC/FEV1 ratio, FEV1 and FVC all greater than the lower limit of normal; mean forced expiratory flow at 25 to 75% of CVF (FEF25-75%) >80% of predicted value and absence of concavity on the forced expiratory flow curve, as evaluated by a trained respirologist; total lung capacity (TLC) greater than the lower limit of normal; residual volume (RV), functional residual capacity (FRC), expiratory reserve volume (ERV), inspiratory capacity (IC) and VR/TLC ratio all >80% predicted value and diffusion capacity of the lung for carbon monoxide (DLCO) >80% predicted value when corrected for hemoglobin level.
* Body mass index (BMI) <30 kg/m2

Exclusion criteria:

• Post-bronchodilator change in FEV1 and FVC of more than 6% and/or 100 ml.

For Non-smokers group:

Inclusion Criteria:

* No history of tobacco-smoking.
* Normal lung function testing, defined as: FVC/FEV1 ratio, FEV1 and FVC all greater than the lower limit of normal; mean forced expiratory flow at 25 to 75% of CVF (FEF25-75%) >80% of predicted value and absence of concavity on the forced expiratory flow curve, as evaluated by a trained respirologist; total lung capacity (TLC) greater than the lower limit of normal; residual volume (RV), functional residual capacity (FRC), expiratory reserve volume (ERV), inspiratory capacity (IC) and VR/TLC ratio all >80% predicted value and diffusion capacity of the lung for carbon monoxide (DLCO) >80% predicted value when corrected for hemoglobin level.
* Body mass index (BMI) <30 kg/m2

Exclusion criteria:

• Post-bronchodilator change in FEV1 and FVC of more than 6% and/or 100 ml.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will include non-obese adults with or without a history of cigarette smoking who performed normal lung function tests.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

PRIMARY OUTCOMES:
AUC-CV>20% values | Immediately after data acquisition
  Density curves with coefficient values >20% will be compared among the two groups of participants

SECONDARY OUTCOMES:
Relationship between AUC-CV>20% values and lung function data | Immediately after data acquisition
  Correlation between AUC-CV>20% values and forced expiratory volume in 1 second, forced vital capacity, residual volume, lung clearance index and diffusion capacity for carbon monoxide
Relationship between AUC-CV>20% values and clinical symptoms | Immediately after data acquisition
  Correlation between AUC-CV>20% values and dyspnea severity (modified medical research council scale) and respiratory symptoms (COPD assessment test)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno-Pierre Dubé, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No